CLINICAL TRIAL: NCT01333111
Title: A Multi-centre, Single-blind Trial Evaluating Safety and Efficacy, Including Pharmacokinetics, of NNC-0156-0000-0009 When Used for Treatment and Prophylaxis of Bleeding Episodes in Patients With Haemophilia B
Brief Title: Safety and Efficacy of NNC-0156-0000-0009 in Haemophilia B Patients
Acronym: paradigm™ 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NN7999-3747; 2010-023069-24 (EudraCT Number); U1111-1119-6415 (Other: WHO); JapicCTI-111644 (Other: Japic)
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Congenital Bleeding Disorder; Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prophylaxis, high dose (trial duration 52 weeks) (Experimental)
  Interventions: Drug: nonacog beta pegol
- Prophylaxis, low dose (trial duration 52 weeks) (Experimental)
  Interventions: Drug: nonacog beta pegol
- On-demand (trial duration 28 weeks) (Experimental)
  Interventions: Drug: nonacog beta pegol

INTERVENTIONS:
Drug: nonacog beta pegol — One single dose administered intravenously (into the vein) once weekly. Patients will receive instruction on how to treat any bleeding episode they may experience
  Other Names: NNC-0156-0000-0009
  Arms: Prophylaxis, high dose (trial duration 52 weeks)
Drug: nonacog beta pegol — One single dose administered intravenously (into the vein) once weekly. Patients will receive instruction on how to treat any bleeding episode they may experience
  Other Names: NNC-0156-0000-0009
  Arms: Prophylaxis, low dose (trial duration 52 weeks)
Drug: nonacog beta pegol — Patients will treat themselves with either a low or a high dose dependent on the severity of the bleeding episode
  Other Names: NNC-0156-0000-0009
  Arms: On-demand (trial duration 28 weeks)

SUMMARY:
This trial is conducted in Africa, Asia, Europe, Japan and North America. The aim of this trial is to evaluate the safety and efficacy, including pharmacokinetics (the rate at which the body eliminates the trial drug), of NNC-0156-0000-0009 (nonacog beta pegol) when used for treatment and prophylaxis of bleeding episodes in patients with haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with moderately severe or severe congenital haemophilia B with a factor IX activity of 2% or below according to medical records
* History of at least 150 exposure days to other factor IX products
* Patients currently treated on-demand with at least 6 bleeding episodes during the last 12 months or at least 3 bleeding episodes during the last 6 months, or patients currently on prophylaxis

Exclusion Criteria:

* Known history of factor IX inhibitors based on existing medical records, laboratory report reviews and patient and legally acceptable representative (LAR) interviews
* HIV (Human immunodeficiency virus) positive, with a viral load equal to or above 400,000 copies/mL and/or CD4+ lymphocyte count equal to or below 200/microL
* Congenital or acquired coagulation disorders other than haemophilia B
* Previous arterial thrombotic events (e.g. myocardial infarction and intracranial thrombosis) or previous deep venous thrombosis or pulmonary embolism (as defined by available medical records)
* Immune modulating or chemotherapeutic medication

Ages: 13 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-04-27 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2013-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (42):
- United States (12):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Houston, Texas
- Novo Nordisk Investigational Site, Edmonton, Alberta, Canada
- France (2):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Lyon
- Germany (4):
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Hanover
- Novo Nordisk Investigational Site, Budapest, Hungary
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Japan (5):
  - Novo Nordisk Investigational Site, Kawasaki-shi, Kanagawa
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Nishinomiya-shi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Suginami-ku, Tokyo
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Utrecht, Netherlands
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Novo Nordisk Investigational Site, Parktown Johannesburg, Gauteng, South Africa
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Kayseri
  - Novo Nordisk Investigational Site, Konya
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Oxford

REFERENCES:
- [Background] Collins PW, Young G, Knobe K, Karim FA, Angchaisuksiri P, Banner C, Gursel T, Mahlangu J, Matsushita T, Mauser-Bunschoten EP, Oldenburg J, Walsh CE, Negrier C; paradigm 2 Investigators. Recombinant long-acting glycoPEGylated factor IX in hemophilia B: a multinational randomized phase 3 trial. Blood. 2014 Dec 18;124(26):3880-6. doi: 10.1182/blood-2014-05-573055. Epub 2014 Sep 26. PMID 25261199
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 40 sites that screened subjects, 39 sites enrolled subjects. The trial was therefore conducted at 39 sites in 13 countries, as follows: France (1); Germany (3); Italy (2); Japan (5); Macedonia (2); Malaysia (1) Netherlands (1); Russia (2); South Africa(1); Thailand (2); Turkey (3); United Kingdom (4) and United States (12).
Groups:
- Prophylaxis, Low Dose 10 U/kg (52 Weeks): Subjects were randomised to either prophylaxis 10 U/kg or 40 U/kg arm. Subjects in this arm received 10 U/kg nonacog beta pegol dose once weekly (every 7th day ± 24 hours) for a period of 52 weeks. Nonacog beta pegol was given as an intravenous bolus injection with the maximum injection rate at 4 mL/min. Mild and moderate bleeding episodes were treated with 40 U/kg. Severe bleeding episodes were treated with 80 U/kg.
- Prophylaxis, High Dose 40 U/kg (52 Weeks): Subjects were randomised to either prophylaxis 10 U/kg or 40 U/kg arm. Subjects in this arm received 40 U/kg nonacog beta pegol dose once weekly (every 7th day ± 24 hours) for a period of 52 weeks. Nonacog beta pegol was given as an intravenous bolus injection with the maximum injection rate at 4 mL/min. Mild and moderate bleeding episodes were treated with 40 U/kg. Severe bleeding episodes were treated with 80 U/kg.
- On-Demand (28 Weeks): Subjects enrolled in this on-demand arm were treated for bleeding episodes on demand with nonacog beta pegol during a period of 28 weeks. Nonacog beta pegol was given as an intravenous bolus injection with the maximum injection rate at 4 mL/min. Mild and moderate bleeding episodes were treated with 40 U/kg. Severe bleeding episodes were treated with 80 U/kg.
Period: Overall Study
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks) | On-Demand (28 Weeks)
Started | 30 | 29 | 15
Completed | 28 | 26 | 13
Not Completed | 2 | 3 | 2
Not completed — patient undergoing major surgery | 0 | 2 | 0
Not completed — personal reasons | 0 | 0 | 1
Not completed — unclassified | 1 | 0 | 0
Not completed — withdrawal criteria | 0 | 1 | 0
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Ineffective therapy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all subjects exposed to nonacog beta pegol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks) | On-Demand (28 Weeks) | Total
Number analyzed (Participants) | 30 | 29 | 15 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (13.9) | 30 (15.8) | 32.4 (12.0) | 31.4 (14.2)
Age, Customized [Number; unit: Participants]
  <=17 years | 7 | 9 | 2 | 18
  18-64 years | 23 | 19 | 13 | 55
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 30 | 29 | 15 | 74

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Inhibitory Antibodies Against Factor IX Defined as Titre Equal to or Above 0.6 BU (Bethesda Units)
Description: Inhibitors were analysed with either the Nijmegen modified factor IX Bethesda assay or a heat/cold Nijmegen modified factor IX Bethesda assay. Number of subjects who developed inhibitory antibodies against factor IX are reported.
Time Frame: 52 weeks after treatment start for patients on prophylaxis
Population: Full analysis set included all subjects exposed to nonacog beta pegol. Subjects in prophylaxis arm were included for this analysis.
Measure: Number; unit: Number of subjects
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks)
Number analyzed (Participants) | 30 | 29
Number of subjects | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Incidence of Inhibitory Antibodies Against Factor IX Defined as Titre Equal to or Above 0.6 BU (Bethesda Units)
Description: as for outcome 1
Time Frame: 28 weeks after treatment start on on-demand treatment
Population: Full analysis set included all subjects exposed to nonacog beta pegol. Subjects in on-demand arm were included for this analysis.
Measure: Number; unit: number of subjects
Arm/Group | On-Demand (28 Weeks)
Number analyzed (Participants) | 15
number of subjects | 0

3. Secondary Outcome: Haemostatic Effect of NNC-0156-0000-0009 When Used for Prophylaxis of Bleeding Episodes, Assessed as Success/Failure Based on a Four-point Scale for Haemostatic Response
Description: Haemostatic response after treatment of a bleed with nonacog beta pegol was evaluated on a 4 point scale as excellent, good, moderate or poor. A success rate was calculated based on counting good or excellent as successes and poor and moderate as failures.
  * Excellent - abrupt pain relief and/or clear improvement in objective signs of bleeding within 8 hours after a single injection
  * Good - noticeable pain relief and/or improvement in signs of bleeding within 8 hours after a single injection
  * Moderate - probable or slight beneficial effect within the first 8 hours after the first injection but requiring more than one injection within 8 hours
  * Poor - no improvement, or worsening of symptoms within 8 hours after two injections.
  The success rate and 95% confidence interval (CI) are reported here.
Time Frame: 52 weeks after treatment start for patients on prophylaxis
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of bleeding episodes
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks)
Number analyzed (Participants) | 30 | 29
percentage of bleeding episodes | 86.9 [76.5 to 93.1] | 97.1 [90.0 to 99.2]

4. Secondary Outcome: Haemostatic Effect of NNC-0156-0000-0009 When Used for Treatment of Bleeding Episodes, Assessed as Success/Failure Based on a Four-point Scale for Haemostatic Response
Description: as for outcome 3
Time Frame: 28 weeks after treatment start on on-demand treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of bleeding episodes
Arm/Group | On-Demand (28 Weeks)
Number analyzed (Participants) | 15
percentage of bleeding episodes | 95.1 [87.0 to 98.2]

5. Secondary Outcome: Number of Bleeding Episodes Per Patient During Routine Prophylaxis
Description: The number of bleeding episodes per patient during routine prophylaxis was assessed using the individual annualised bleeding rates (spontaneous and traumatic bleeding episodes per patient per year).
Time Frame: 52 weeks after treatment start for patients on prophylaxis
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: bleeds/patient/year
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks)
Number analyzed (Participants) | 30 | 29
bleeds/patient/year | 2.93 (5.41) [0.99 to 6.02] | 1.04 (7.41) [0.00 to 4.00]

6. Secondary Outcome: Factor IX Trough Levels
Description: The mean pre-dose factor IX levels was measured with the one-stage clotting assay during the trial. Lowest factor IX activity recorded during single-dose and steady state, immediately before next dose was given. The analysis was based on a mixed model on the log-transformed plasma factor IX activity with subject as a random effect. The estimated mean factor IX trough level was presented back-transformed to the natural scale.
Time Frame: 52 weeks after treatment start for patients on prophylaxis
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks)
Number analyzed (Participants) | 30 | 29
U/mL | 0.085 [0.077 to 0.093] | 0.273 [0.248 to 0.300]

7. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: The incidence of adverse events were summarised by the rate of AEs (number of AEs per patient years of exposure [PYE]). Number of adverse events per PYE is number of adverse events /total time in trial. All adverse events reported are treatment emergent (any adverse events which occurred after trial product administration).
Time Frame: at 56 weeks ±2 weeks for patients on prophylaxis
Population: Safety analysis set included all subjects exposed to nonacog beta pegol. Subjects in prophylaxis arm were included for this analysis.
Measure: Number; unit: number of AEs per PYE
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks)
Number analyzed (Participants) | 30 | 29
number of AEs per PYE | 2.62 | 3.83

8. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: The incidence of adverse events were summarised by the rate of AEs (number of AEs per PYE). Number of adverse events per PYE is number of adverse events /total time in trial. All adverse events reported are treatment emergent (any adverse events which occurred after trial product administration).
Time Frame: at 32 weeks ±2 weeks for patients on on-demand treatment
Population: Safety analysis set included all subjects exposed to nonacog beta pegol.Subjects in on-demand arm were included for this analysis.
Measure: Number; unit: number of AEs per PYE
Arm/Group | On-Demand (28 Weeks)
Number analyzed (Participants) | 15
number of AEs per PYE | 4.14

9. Secondary Outcome: Incidence of Serious Adverse Events (SAEs)
Description: SAE was defined as an AE that resulted in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect. The incidence of SAEs were summarised by the rate of SAEs (number of SAEs per PYE). Number of SAEs per PYE is number of SAEs/total time in trial. All SAEs reported are treatment emergent (any serious adverse events which occurred after trial product administration).
Time Frame: at 56 weeks ±2 weeks for patients on prophylaxis
Population: as for outcome 7
Measure: Number; unit: number of SAEs per PYE
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks)
Number analyzed (Participants) | 30 | 29
number of SAEs per PYE | 0.03 | 0.11

10. Secondary Outcome: Incidence of Serious Adverse Events (SAEs)
Description: as for outcome 9
Time Frame: at 32 weeks ±2 weeks for patients on on-demand treatment
Population: Safety analysis set included all subjects exposed to nonacog beta pegol. Subjects in on-demand arm were included for this analysis.
Measure: Number; unit: number of SAEs per PYE
Arm/Group | On-Demand (28 Weeks)
Number analyzed (Participants) | 15
number of SAEs per PYE | 0

11. Secondary Outcome: Host Cell Proteins (HCP) Antibodies
Description: Subjects who were positive for anti-Host Cell Protein (HCP) antibodies.
Time Frame: 52 weeks after treatment start for patients on prophylaxis
Population: as for outcome 7
Measure: Number; unit: number of subjects
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks)
Number analyzed (Participants) | 30 | 29
number of subjects | 0 | 1

12. Secondary Outcome: Host Cell Proteins (HCP) Antibodies
Description: Subjects who were positive for anti-HCP antibodies.
Time Frame: 28 weeks after treatment start on on-demand treatment
Population: as for outcome 10
Measure: Number; unit: number of subjects
Arm/Group | On-Demand (28 Weeks)
Number analyzed (Participants) | 15
number of subjects | 0

ADVERSE EVENTS:
Time Frame: For the subjects treated with prophylaxis, adverse events were assessed for 52 weeks + 4 weeks. For the subjects treated on-demand, adverse events were assessed for 28 weeks + 4 weeks.
Description: Treatment-emergent adverse events were defined as any adverse events which occurred after trial product administration. Analysis was based on the safety analysis set.
Arm/Group | Prophylaxis, Low Dose 10 U/kg (52 Weeks) | Prophylaxis, High Dose 40 U/kg (52 Weeks) | On-Demand (28 Weeks)
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/29 | 0/15
Other Adverse Events (participants affected / at risk) | 21/30 | 19/29 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis, Low Dose 10 U/kg (52 Weeks) (N=30) | Prophylaxis, High Dose 40 U/kg (52 Weeks) (N=29) | On-Demand (28 Weeks) (N=15)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis, Low Dose 10 U/kg (52 Weeks) (N=30) | Prophylaxis, High Dose 40 U/kg (52 Weeks) (N=29) | On-Demand (28 Weeks) (N=15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (2)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (7) | 2 (3)
Influenza (Infections and infestations) | 4 (4) | 3 (5) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (9) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Prothrombin level increased (Investigations) | 0 (0) | 2 (4) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 2 (4) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder developmental (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.